CLINICAL TRIAL: NCT02999269
Title: ECT Pulse Amplitude and Medial Temporal Lobe Engagement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: The Mind Research Network (Other); University of Texas (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christopher Abbott, Medical Director ECT Service, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5U01MH111826 (NIH); 5U01MH111826 (NIH)
Record Dates: First submitted 2016-08-16; First posted 2016-12-21 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Major Depressive Disorder
Keywords: electroconvulsive therapy; MRI; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Subjects randomized to right unilateral ECT with 600, 700, or 800 mA pulse amplitude.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (participant and outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 600 mA Right Unilateral ECT (Experimental): MECTA Spectrum 5000Q Amplitude
  Interventions: Device: MECTA Spectrum 5000Q Amplitude
- 700 mA Right Unilateral ECT (Experimental): MECTA Spectrum 5000Q Amplitude
  Interventions: Device: MECTA Spectrum 5000Q Amplitude
- 800 mA Right Unilateral ECT (Active Comparator): MECTA Spectrum 5000Q Amplitude
  Interventions: Device: MECTA Spectrum 5000Q Amplitude

INTERVENTIONS:
Device: MECTA Spectrum 5000Q Amplitude — Current

SUMMARY:
Electroconvulsive therapy (ECT) remains the gold-standard treatment for patients with depressive episodes. During a typical four-week ECT series, most depressive episodes will respond to treatment and people will improve their level of functioning (return to work or family). Independent of the antidepressant effect of ECT, many patients experience transient memory impairment. This investigation will examine the impact of one ECT parameter (pulse amplitude or current) on brain changes (structure of connections within the brain) and clinical outcomes. The goal of this investigation is to determine the optimal parameter for an individual patient that will maintain the clinical response (reduce depression severity) and minimize side effects (eliminate memory issues related to treatment).

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) remains the gold-standard treatment for patients with depressive episodes. During a typical four-week ECT series, most depressive episodes remit, and formerly suicidal or psychotically depressed patients will resume their premorbid levels of functioning. Independent of the antidepressant effect of ECT, many patients experience debilitating but transient cognitive effects such as attention and memory deficits. These unwanted side effects are particularly troubling for older patients who are more likely to have existing cognitive deficits. Both the stimulus delivery (electrode placement, pulse amplitude, and pulse width) and seizure induction appear to work in synergy, but the underlying mechanism of action for successful response has yet to be fully elucidated. Moreover, further work is needed to understand the relationship between clinical improvement and cognitive impairment. This investigation will examine the clinical and neurocognitive impact of targeted medial temporal lobe engagement as a function of pulse amplitude, one of several variable factors influencing the ECT charge. The ECT charge is measured in millicoulombs (mC) and derived from multiplying pulse train duration, pulse-pair frequency, pulse width, and pulse amplitude. Pulse amplitude determines the induced electric field strength in the brain and is presently fixed at 900 milliamperes (mA) with no clinical or scientific justification. The central hypothesis of this investigation is that the optimal pulse amplitude for an individual patient will enhance neuroplasticity (clinical response) while minimizing the disruption of dominant hemisphere hippocampal cognitive circuitry (resulting in cognitive stability). The preliminary data informs the dosage range between 600 and 800 mA. Pulse amplitudes outside of this range compromise efficacy (500 mA) or may increase risk of cognitive impairment (900 mA). The first aim of this investigation will identify the electric field strength and neuroplasticity associated with clinical response. Critically, this aim will establish the neuroplasticity threshold, which is defined as the electric field strength necessary to induce neuroplasticity. The second aim will detect the neural correlates of ECT-mediated cognitive changes, which may be related to disrupted dominant hemisphere long-term potentiation. The third aim will use data-driven dual regression to predict the optimal pulse amplitude for an individual patient. This contribution will be significant because the electric field, when manipulated by pulse amplitude, can subsequently maximize hippocampal neuroplasticity (efficacy) and minimize disrupted connectivity (cognitive stability) thus improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of major depressive disorder (with or without psychotic features)
2. the clinical indications for ECT including treatment resistance or a need for a rapid and definitive response
3. Hamilton Depression Rating Scale 24-item (HDRS-24) > 21
4. age range between 50 and 80 years of age
5. right-handedness

Exclusion Criteria:

1. Defined neurological or neurodegenerative disorder (e.g., history of head injury with loss of consciousness > 5 minutes, epilepsy, Alzheimer's disease)
2. other psychiatric conditions (e.g., schizophrenia, schizoaffective disorder, bipolar disorder)
3. current drug or alcohol use disorder, except for nicotine; and 4) contraindications to MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Abbott, MD, Principal Investigator — University of New Mexico
Locations (1):
- Chris Abbott, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
National Data Archive (NDA)
Supporting Information: Study Protocol
Time Frame: Clinical, cognitive and MRI data was uploaded to NDA.
Access Criteria: per NDA protocol

REFERENCES:
- [Result] Abbott CC, Quinn D, Miller J, Ye E, Iqbal S, Lloyd M, Jones TR, Upston J, Deng Z, Erhardt E, McClintock SM. Electroconvulsive Therapy Pulse Amplitude and Clinical Outcomes. Am J Geriatr Psychiatry. 2021 Feb;29(2):166-178. doi: 10.1016/j.jagp.2020.06.008. Epub 2020 Jun 17. PMID 32651051
- [Derived] Qi S, Calhoun VD, Zhang D, Miller J, Deng ZD, Narr KL, Sheline Y, McClintock SM, Jiang R, Yang X, Upston J, Jones T, Sui J, Abbott CC. Links between electroconvulsive therapy responsive and cognitive impairment multimodal brain networks in late-life major depressive disorder. BMC Med. 2022 Dec 8;20(1):477. doi: 10.1186/s12916-022-02678-6. PMID 36482369

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 600 mA Right Unilateral ECT | 700 mA Right Unilateral ECT | 800 mA Right Unilateral ECT
Started | 20 | 20 | 20
Completed | 16 | 15 | 16
Not Completed | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mA Right Unilateral ECT | 700 mA Right Unilateral ECT | 800 mA Right Unilateral ECT | Total
Number analyzed (Participants) | 16 | 15 | 16 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 8 | 7 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8) | 64 (7) | 67 (10) | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 11 | 32
  Male | 4 | 6 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 15
  Not Hispanic or Latino | 11 | 10 | 11 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 15 | 14 | 15 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Hamilton Depression Rating Scale - 24 items Clinician rated measure of depression severity, range 0 -76 with higher scores indicating more severe depression
  participants
    United States | 16 | 15 | 16 | 47
Hamilton Depression Rating Scale 24 items [Mean (Standard Deviation); unit: units on a scale] — Clinician rated scale obtained during structured interview with subject. The scoring range is from 0 to 76 with higher scores indicating more depression severity
  units on a scale | 37.0 (7.8) | 38.0 (7.5) | 33.8 (6.7) | 36.3 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Hamilton Depression Rating Scale - 24 item. Scores range from 0 to 76 (higher scores indicate more depression severity)
Time Frame: post-ECT Hamilton Depression Rating Scale -24 item. The time frame is 4 weeks after study initiation.
Population: full longitudinal model with an unstructured repeated measures covariance matrix
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 600 mA Right Unilateral ECT | 700 mA Right Unilateral ECT | 800 mA Right Unilateral ECT
Number analyzed (Participants) | 16 | 15 | 16
score on a scale | 22.5 (2.3) | 12.0 (2.1) | 14.1 (2.4)
Statistical Analysis 1: Comparison: 600 mA Right Unilateral ECT vs 700 mA Right Unilateral ECT vs 800 mA Right Unilateral ECT; For the primary outcomes (change in HDRS24), we performed a full longitudinal model with an unstructured repeated measures covariance matrix on subjects who completed the study in the assigned treatment arm. The dependent variable was HDRS at each visit and the independent variables included progress (time within the ECT series: pre-, mid-, and post-ECT), amplitude, age, sex, pulse width and the following interactions: progress/amplitude, progress/sex, and progress/pulse width; Test type: Superiority; p = 0.04, Regression, Linear — p-value for time by amplitude interaction; Time-by-amplitude interaction (F4, 72 = 2.65, p = 0.04)
Statistical Analysis 2: Comparison: 600 mA Right Unilateral ECT vs 700 mA Right Unilateral ECT vs 800 mA Right Unilateral ECT; Test type: Superiority; p = 0.0001, Regression, Linear

2. Primary Outcome: Cognition
Description: Hopkins Verbal Learning Trial-Revised (percent retention score, range 0 - 100, higher is better)
Time Frame: post-ECT Hopkins Verbal Learning Trial-Revised (percent retention score, range 0 - 100, higher is better). The time frame is 4 weeks after study initiation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 600 mA Right Unilateral ECT | 700 mA Right Unilateral ECT | 800 mA Right Unilateral ECT
Number analyzed (Participants) | 16 | 15 | 16
score on a scale | 57.3 (10) | 68 (9) | 62 (10)
Statistical Analysis 1: Comparison: 600 mA Right Unilateral ECT vs 700 mA Right Unilateral ECT vs 800 mA Right Unilateral ECT; Test type: Superiority; p = 0.37, Regression, Linear
Statistical Analysis 2: Comparison: 600 mA Right Unilateral ECT vs 700 mA Right Unilateral ECT vs 800 mA Right Unilateral ECT; Test type: Superiority; p = 0.50, Regression, Linear — p-value is time-by-amplitude interaction
Statistical Analysis 3: Comparison: 600 mA Right Unilateral ECT vs 700 mA Right Unilateral ECT vs 800 mA Right Unilateral ECT; Test type: Superiority; p < 0.01, Regression, Linear — Progress (F2,71 = 11.15, p < 0.01)

ADVERSE EVENTS:
Time Frame: Each subject was evaluated for adverse effects over the 4-week study protocol.
Arm/Group | 600 mA Right Unilateral ECT | 700 mA Right Unilateral ECT | 800 mA Right Unilateral ECT
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 6/20 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mA Right Unilateral ECT (N=20) | 700 mA Right Unilateral ECT (N=20) | 800 mA Right Unilateral ECT (N=20)
headache (Nervous system disorders) | 5 (10) | 6 (17) | 6 (17) — post-procedure headache, all cases resolved with over the counter medications (Tylenol)

LIMITATIONS AND CAVEATS:
Subjects discontinued scheduled antidepressant and antipsychotic medications prior to the first imaging assessment, but as-needed medications (lorazepam, quetiapine, trazodone) were permissible with dose restrictions during the ECT series. Second, our study design included a change in pulse width (from 0.3 to 1.0 ms). Each amplitude arm had a very limited number of subjects with brief pulse width. The relationship between amplitude and pulse width will require more research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02999269/Prot_SAP_000.pdf